CLINICAL TRIAL: NCT05275894
Title: Non-surgical Treatment of Peri-implantitis With Electrolytic Cleaning: a Pilot Study
Brief Title: Non-surgical Electrolytic Cleaning Peri-implantitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCM ACA
Record Dates: First submitted 2022-02-02; First posted 2022-03-11 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-10

CONDITIONS: Peri-Implantitis
Keywords: Peri-implantitis; Electrolytic cleaning; Implant decontamination; Non-surgical treatment
MeSH Terms: conditions — Peri-Implantitis | interventions — Microsurgery; Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-surgical electrolytic cleaning (Experimental): * Implant hygiene instructions and removal of the prosthesis
  * Local anaesthesia
  * Removal of the granulation tissue and mucosa and bone defect curettage with a steel curette 4R/4L (Hu-Friedy, Chicago, IL, USA)
  * Removal of supra and submucosal calculus with slim ultrasonic devices (Piezon PS instrument EMS; Nyon, Swiss).
  * Erythritol air powder-spray system (Air-flow ® master piezon, EMS, Nyon swiss) implant surface treatment. This will be performed by separating the soft tissue with the aim of a periodontal probe (CP 15, Hu-Friedy, Chicago, IL, USA).
  * Electrolytic cleaning of the implant surface following manufacturer's instructions (GalvoSurge Dental AG, Widnau, Switzerland), with the help of a non-metal periodontal probe to separate the soft tissues and aim the implant surface in all its length.
  * Antibiotic treatment (Metronidazole 500 mg, every day/ 7 day).
  * If necessary, modification and polishing of the prosthesis to make it cleanable.
  Interventions: Behavioral: Implant hygiene instructions and removal of the prosthesis; Procedure: Non-surgical peri-implantitis treatment /microsurgery; Procedure: Implant surface decontamination 1(ultrasonic device); Procedure: Implant surface decontamination 2 (air polishing); Procedure: Implant surface decontamination 3 (electrolytic cleaning); Drug: Antibiotic treatment (Metronidazole); Procedure: Modification and polishing of the prosthesis

INTERVENTIONS:
Behavioral: Implant hygiene instructions and removal of the prosthesis — Verbal instructions on implant hygiene practices and removal of the implant supported prosthesis
Procedure: Non-surgical peri-implantitis treatment /microsurgery — Removal of the granulation tissue and mucosa and bone defect curettage with a steel curette 4R/4L (Hu-Friedy, Chicago, IL, USA) after applying local anestesia
Procedure: Implant surface decontamination 1(ultrasonic device) — Removal of supra and submucosal calculus with slim ultrasonic devices (Piezon PS instrument EMS; Nyon, Swiss).
Procedure: Implant surface decontamination 2 (air polishing) — Erythritol air powder-spray system (Air-flow ® master piezon, EMS, Nyon swiss) implant surface treatment. This will be performed by separating the soft tissue with the aim of a periodontal probe (CP 15, Hu-Friedy, Chicago, IL, USA).
Procedure: Implant surface decontamination 3 (electrolytic cleaning) — Electrolytic cleaning of the implant surface following manufacturer's instructions (GalvoSurge Dental AG, Widnau, Switzerland), with the help of a non-metal periodontal probe to separate the soft tissues and aim the implant surface in all its length.
Drug: Antibiotic treatment (Metronidazole) — Antibiotic treatment (Metronidazole 500 mg, every day/ 7 day).
  Other Names: Metronidazole
Procedure: Modification and polishing of the prosthesis — If necessary, modification and polishing of the prosthesis to make it cleanable.

SUMMARY:
Electrolytic cleaning is a promising treatment for dental implant decontamination, but this mode of therapy has not yet been clinically tested as an adjunct to the non-surgical treatment of periimplantitis.

A prospective clinical and radiographic case series study will be performed to evaluate the clinical performance of the adjunctive use of electrolytic cleaning as an adjunct to a non-surgical therapy protocol that includes curettage of the peri-implant soft tissue. This is study is a proof of principle study, thus, a case series study is selected to start with. If the results of this case series study are favourable, a future study with a clinical trial design is then planned to do.

DETAILED DESCRIPTION:
Electrolytic cleaning is a promising treatment for dental implant decontamination, but this mode of therapy has not yet been clinically tested as an adjunct to the non-surgical treatment of periimplantitis. Electrolytic cleaning is a promising treatment for dental implant decontamination, but this mode of therapy has not yet been clinically tested as an adjunct to the non-surgical treatment of periimplantitis.This is study is a proof of principle study, thus, a case series study is selected to start with. As this is a pilot study to test for the first time the electrolytic cleaning under non-surgical therapy, the sample size has been estimated in a minimum of 25 patients. If the results of this case series study are favourable, a future study with a clinical trial design is then planned to do.

Therapeutic success is defined as as a composite index (Sanz & Chapple 2012 criteria of disease resolution) that includes: (1) probing pocket depth < 5 mm, (2) no bleeding on probing/suppuration and (3) no additional bone loss, at 6 and 12 months). Secondary objectives are: Changes in the clinical outcomes measurements.Changes in the radiological outcomes measurements. Changes in the patient-reported outcomes (PROMs). Evaluation of the outcomes related to the prosthetic restoration.

This study will be carried out in the following centers:

* Postgraduate Periodontal Clinic at the Faculty of Odontology-Universidad Complutense of Madrid (Spain)
* CEOSA-Madrid Private Dental Centre

After the non-surgical therapy, patients will be recalled for control visits, with supra- gingival removal of biofilm with air polishing without anaesthesia at:

* 3 months.
* 6 months.
* 12 months. After non-surgical therapy, patients will be included in a strict peri-implant maintenance therapy program to avoid re-contamination of the affected implants. Removal of biofilm with air polishing without anaesthesia and oral hygiene instruction reinforcement will be performed at: 3 months, 6 months, 9 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age > 18 years.
* Presence of at least 1 implant with the diagnose of peri-implantitis (Berglundh et al. 2018; Renvert et al. 2018)
* Peri-implant bone loss < 2/3
* History of treated periodontal diseases (Caton 2018).
* Screw retained prosthesis that can be easily unscrewed.
* Prosthesis that allows access to biofilm control by the patient, or which can be modified accordingly.
* Absence of implant mobility

Exclusion Criteria:

Systemic exclusion criteria

* Pregnant or lactating women Non-surgical electrolytic cleaning CONFIDENTIAL
* Patients chronically treated (i.e., two weeks or more) with any medication known to affect periodontal/peri-implant status (i.e., antibiotics intake within 3 months prior to the initiation)
* Medical conditions requiring prolonged use of steroids and/or with medications that could interfere with bone metabolism.
* History of leukocyte dysfunction and deficiencies.
* History of neoplastic disease requiring the use of radiation or chemotherapy.
* Patients with chronic renal failure requiring dialysis.
* Patients with metabolic bone disorders such as osteoporosis treated with antiresoptive medications.
* History of uncontrolled endocrine disorders: hypothyroidism or diabetes.
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene or patients unable to use daily interproximal cleaning.
* Alcoholism or drug abuse.
* History of immunodeficiency syndromes.
* Tobacco consumption (smoking more than 10 cigarettes per day)
* Conditions or circumstances, which in the opinion of the investigator, would avoid the completion of study participation, or interfere with analysis of study results, such as history of non-compliance or unreliability, or do have any additional medical condition that contraindicates non-surgical treatment

Local exclusion criteria

* Mucosal diseases such as erosive lichen planus in the area to be treated.
* History of local irradiation therapy.
* Implants with peri-implant bone loss beyond 2/3 of the implant length

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Peri-implant disease resolution at 6 month | 6 months
  Probing depth < 5 mm, with absence of bleeding or suppuration and no additional bone loss (Sanz & Chapple 2012)
Peri-implant disease resolution at 12 month | 12 months
  Probing depth < 5 mm, with absence of bleeding or suppuration and no additional

SECONDARY OUTCOMES:
Implant survival rate at 6 months | 6 months
  Survival of installed implants as defined by Misch et al., 2007: presence in the mouth, no mobility, no pain upon function, radiographic bone loss less than 1⁄2, no uncontrolled infection.
Implant survival rate at 12 months | 12 months
  Survival of installed implants as defined by Misch et al., 2007: presence in the mouth, no mobility, no pain upon function, radiographic bone loss less than 1⁄2, no uncontrolled infection.
Implant plaque index at 6 months | 6 months
  Implant plaque index (PI) (at 6 sites/implant)(+/-).
Implant plaque index at 12 months | 12 months
  Implant plaque index (PI) (at 6 sites/implant)(+/-).
Peri-implant probing depth at 6 months | 6 months
  Peri-implant probing depth (PD) (at 6 sites/implant) recorded using a CPC-15 periodontal probe at 6 sites/implant (Hu-Friedy, Leinmen, Germany).
Peri-implant probing depth at 12 months | 12 months
  Peri-implant probing depth (PD) (at 6 sites/implant) recorded using a CPC-15 periodontal probe at 6 sites/implant (Hu-Friedy, Leinmen, Germany).
Bleeding on probing at 6 months | 6 months
  Bleeding on probing (BOP) from the peri-implant mucosa (measured at 6 sites/implant) (+/-).
Bleeding on probing at 12 months | 12 months
  Bleeding on probing (BOP) from the peri-implant mucosa (measured at 6 sites/implant) (+/-).
Suppuration at 6 months | 6 months
  Presence or absence of suppuration from the peri-implant mucosa (measured at 6 sites/implant) (+/-) nice, regular, unpleasant, very unpleasant).
Suppuration at 12 months | 12 months
  Presence or absence of suppuration from the peri-implant mucosa (measured at 6 sites/implant) (+/-)
Recession of the mucosal margin at 6 months | 6 months
  Recession of the mucosal margin, keratinized mucosa (at 6 sites/implant) (+/-).recorded using a CPC-15 periodontal probe at 6 sites/implant (Hu-Friedy, Leinmen, Germany).
Recession of the mucosal margin at 12 months | 12 months
  Recession of the mucosal margin, keratinized mucosa (at 6 sites/implant) (+/-).recorded using a CPC-15 periodontal probe at 6 sites/implant (Hu-Friedy, Leinmen, Germany).
Bone loss at 6 months | 6 months
  Distance between bone crest and implant shoulder at mesial and distal site. For standardization of the periapical radiographs the same film holder-beam aiming device will be applied to each treated implant (i.e. Rinn System, RWT window x-ray system or Non-surgical electrolytic cleaning CONFIDENTIAL similar). The radiographs will be taken with the film placed parallel to the implants and the x-ray beam directed perpendicular to the implants. The quality/contrast should be good enough to clearly identify the complete implant and its essential structures.
  Digital radiographs will be evaluated using a software (OsiriX Imaging Software, Pixmeo, Geneva, Switzerland) calibrating the distances with implant wide and length.
Bone loss at 12 months | 12 months
  Distance between bone crest and implant shoulder at mesial and distal site. For standardization of the periapical radiographs the same film holder-beam aiming device will be applied to each treated implant (i.e. Rinn System, RWT window x-ray system or Non-surgical electrolytic cleaning CONFIDENTIAL similar). The radiographs will be taken with the film placed parallel to the implants and the x-ray beam directed perpendicular to the implants. The quality/contrast should be good enough to clearly identify the complete implant and its essential structures.
  Digital radiographs will be evaluated using a software (OsiriX Imaging Software, Pixmeo, Geneva, Switzerland) calibrating the distances with implant wide and length.
Patient centred outcomes of the electrolytic cleaning after 6 months | 6 months
  Patient centred outcomes of the electrolytic cleaning with a 5 options semi-quantitative scale (very nice, nice, regular, unpleasant, very unpleasant).
Patient centred outcomes of the electrolytic cleaning after 12 months | 12 months
  Patient centred outcomes of the electrolytic cleaning with a 5 options semi-quantitative scale (very nice, nice, regular, unpleasant, very unpleasant).
Overall satisfaction after 6 months | 6 months
  Overall satisfaction on a 5 options semi-quantitative scale (very nice, nice, regular, unpleasant, very unpleasant).
Overall satisfaction after 12 months | 12 months
  Overall satisfaction on a 5 options semi-quantitative scale (very nice, nice, regular, unpleasant, very unpleasant).

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz Alonso, Principal Investigator — University Complutense Madrid
Locations (1):
- Ana Carrillo de Albornoz, Madrid, Spain